CLINICAL TRIAL: NCT05850442
Title: The Relationship Between Fibromyalgia Syndrome Parameters With Disease Severity, Pain and the Quality Of Life
Brief Title: The Relationship Between Fibromyalgia Syndrome Parameters With Disease-Pain Severity and the Quality Of Life
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Özlem Kaleoğlu, MD, Principle Investigator, Umraniye Education and Research Hospital
Other Study IDs: B.10.1.THK.4.34.H.GP.0.01/121
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia Syndrome; Anxiety Disorders; Depressive Disorder
MeSH Terms: conditions — Fibromyalgia; Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- FIBROMIYALGIA GROUP: Patients aged between 18-65 who are diagnosed as FMS according to AACR 2016 criterias willing to take part in the study.
  Interventions: Diagnostic Test: Questionary

INTERVENTIONS:
Diagnostic Test: Questionary — Patients will be asked to fill Fibromyalgia Impact Questionary, WHO Short Quality of Life Questionary, McGill Pain Questionary and Beck Anxiety Questionary

SUMMARY:
In this study, the investigators aim to evaluate the relationship between disease severity, quality of life, anxiety and pain level in patients diagnosed with Fibromyalgia Syndrome (FMS) with the parameters according to the American College of Rheumatology (ACR) 2016 diagnostic criteria. According to the 2016 ACR diagnostic criteria, there are 2 separate scales: Widespread Pain Index (WPI) and Symptom Severity (SS) . The relationship between these 2 parameters and the Fibromyalgia Impact Questionnaire, the World Health Organization Short Quality of Life Questionnaire, and the McGill Melzack Pain Questionnaire and Beck Anxiety Questionnaire will be examined.

DETAILED DESCRIPTION:
The aim of this study is to observe the relationship between the WPI and SS parameters in the ACR 2016 criteria for fibromyalgia, separately, with the severity of the disease, pain level, quality of life and anxiety level. Accordingly, the investigators aim to evaluate whether WPI or SS has priority in assessing the severity of the disease. There is no study in the literature comparing the importance of the 2016 ACR diagnostic parameters on the disease effect. In this context, this study will be the first study in the literature and will be very valuable. Patients visiting the outpatient clinic with FMS diagnosis will be evaluated. Patients will be asked to fill the World Health Organization Short Quality of Life Questionnaire, and the McGill Melzack Pain Questionnaire and Beck Anxiety Questionnaire . The patients will be assed by an experienced Physical Medicine and Rehabilitation specialist for SS and WPI scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as FMS according to ACR 2016 criterias

Exclusion Criteria:

* History of Malignity
* History of Rheumatological Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with FMS according to ACR 2016 criteria
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Widespread Pain Index Score | at the start of the study
  Widespread Pain Index Score, Ranging from 0-19. Higher scores mean higher pain scores.
Symptom Severity Score | at the start of the study
  Symptom Severity Score. Ranging from 0-12. Higher scores mean higher symptom scores.

SECONDARY OUTCOMES:
Beck Anxiety Score | at the start of the study
  Beck Anxiety Score, Ranging from 0-63. Higher scores mean anxiety getting worse.
WHO Short Quality of Life Score | at the start of the study
  WHO Short Quality of Life Score, Ranging from 0-100. Higher scores mean better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Özlem Kaleoğlu, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No